CLINICAL TRIAL: NCT00402948
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups, To Evaluate And Compare The Safety, Tolerability And Efficacy Of Two Dosages Of Inhaled TPI ASM8 Administered For 14 Days In Patients With Mild to Moderate Asthma.
Brief Title: Safety and Efficacy of Two Dosages of Inhaled TPI ASM8 Compared to Placebo in Mild to Moderate Asthmatic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of substantial enrollment
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPI ASM8 -204
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: High eosinophils level in sputum
MeSH Terms: conditions — Asthma | interventions — TPI ASM8

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPI ASM8 (Experimental): ASM8 0.25mg
  Interventions: Drug: TPI ASM8
- ASM8 as TPI ASM8 (Experimental): TPI ASM8 0.5mg
  Interventions: Drug: ASM8

INTERVENTIONS:
Drug: TPI ASM8 — 0.25mg, 0.5mg for 14 days, daily dosage
  Arms: TPI ASM8
Drug: ASM8 — inhalation 0.25mg daily for 14 days
  Arms: ASM8 as TPI ASM8

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of two dosages of a new drug TPI ASM8 administered by inhalation for 14 days to mild to moderate asthmatic patients, aged between 18-65, non-smokers . The study will also look at the nature and quantity of inflammatory white cells in the lung secretions and in the blood, and some additional inflammation markers.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 y. old, non or ex-smokers for > 6 months
* Mild to moderate asthmatic in general good health
* On either low-dose inhaled corticosteroid or steroid naive
* No other asthma medication
* Regular sputum producer
* EOS more than 3% at randomization,
* FEV1 > 70%

Exclusion Criteria:

* Respiratory infection within last 4 weeks
* Any condition that may affect the conduct of the study as per the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophils at Day 1 and Day 14 and safety on Day 14 | Prospective

SECONDARY OUTCOMES:
FEV 1 on Day 1 and Day 14 | Prospective
Rescue Medication (albuterol)for 21 days | Prospective
Gene expression ( mRNA, beta-chain and CCR3 on surface receptors of IL-3, IL-5 and GM-CSF | Prospective
Blood eosinophils at Day 0 and Day 15 | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaram Nair, MD, Principal Investigator — Firestone Institute for Respiratory Health
Locations (10):
- Canada (10):
  - Calgary COPD & Asthma Program, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - St-Paul's Hospital, Vancouver, British Columbia
  - McMaster University Hospital, Hamilton, Ontario
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Institut Thoracique de Montreal, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
  - Hopital Laval- Centre de recherche de Cardiologie et Pneumologie, Québec, Quebec